CLINICAL TRIAL: NCT05169671
Title: A Randomized, Placebo-Controlled, Double-Blinded, First-in-Human, Adaptive Study to Evaluate Safety, Tolerability, and Pharmacokinetics of Single Ascending Doses (Part A) and Multiple Ascending Doses (Part B) of Orally Administered ATH-1020 in Healthy Young and Elderly Subjects
Brief Title: Safety, Tolerability, and Pharmacokinetics Study of ATH-1020
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Athira Pharma (Industry)
Collaborators: Biotrial Inc. (Unknown); Alturas Analytics, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATH-1020-0101
Record Dates: First submitted 2021-12-06; First posted 2021-12-27 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Healthy Volunteers
Keywords: Pharmacokinetics; HGF/MET

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ATH-1020 (Experimental): ATH-1020 in oral form. Participants in the single ascending dose cohort (Cohort A) will receive a single dose of ATH-1020. Participants in the multiple ascending dose cohort (Cohort B) will receive up to nine doses of ATH-1020 (up to 4 for cohort B5).
  Interventions: Drug: ATH-1020
- Placebo (Placebo Comparator): Placebo in oral form. Participants in the single ascending dose cohort (Cohort A) will receive a single dose of Placebo. Participants in the multiple ascending dose cohort (Cohort B) will receive up to nine doses of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ATH-1020 — ATH-1020 in oral capsule form
  Arms: ATH-1020
Drug: Placebo — Placebo in oral capsule form
  Arms: Placebo

SUMMARY:
This Phase 1 randomized, placebo-controlled, double-blinded, first-in-human study will evaluate safety, tolerability, and pharmacokinetics of single and multiple ascending doses of ATH-1020 in healthy young and elderly subjects.

DETAILED DESCRIPTION:
This is a Phase 1 first-in-human, 2-part adaptive study. Both Part A and Part B will be performed in a randomized, placebo-controlled, and double-blind manner.

Part A - Single Ascending Dose (SAD) Part A will be a SAD study investigating multiple dose levels of ATH 1020.

Part B - Multiple Ascending Dose (MAD) Part B will be a multiple ascending dose (MAD) study investigating multiple dose levels of ATH-1020.

Subjects in Cohort B5 (4 subjects) will additionally undergo CSF sampling pre-dose on Day 4 and up to 3 post dose timepoints to evaluate ATH-1020 blood-brain-barrier penetration

ELIGIBILITY:
Inclusion Criteria:

All Subjects

1. Body mass index (BMI) of ≥ 18.0 and ≤ 32.0 kg/m2 at Screening, with minimum weight of 60 kg.
2. Subjects in generally good health per the investigator's discretion.
3. Male subjects and their partners must be willing to comply with the contraceptive requirements of the study.
4. Subjects must have adequate venous access.

   Part A (SAD)
5. Male subjects aged 18 to 50 years at the time of signing the informed consent.

   Part B (MAD)
6. Male subjects aged 18 to 50 years (Cohorts B1, B2, B3, and B5); male and post-menopausal female subjects aged 65 to 85 years (Cohort B4) at the time of signing the informed consent.

Exclusion Criteria:

1. History of significant drug allergies (including to any excipients) or of anaphylactic reaction.
2. Any condition per the investigator's discretion, which while not requiring chronic medication use, is likely to require intermittent/acute therapeutic intervention.
3. Any history of seizures or loss of consciousness for an unknown reason.
4. History of or positive results of serology screening for hepatitis B, hepatitis C or human immunodeficiency virus (HIV).
5. Abnormal liver tests
6. Impaired renal function.
7. History of having taken another investigational drug within 30 days prior to Admission (Day -1).
8. Major surgery within 90 days prior to Admission (Day -1) or anticipated surgery during the study.

   Part A (SAD)
9. Female subjects are not permitted.
10. Any medical condition that requires chronic medication use.

    Part B (MAD)
11. A history of intermittent benzodiazepine (short-acting only) or other treatments for insomnia and anxiety are allowed, provided that the subject is able to abstain from their use during the Screening period, and from Admission until discharge from the study.
12. Reported changes in cognition and reported history of declines in everyday life in the last year.

    Part B (MAD) CSF Sampling (Cohort B5)
13. Subject history of or current contraindication to lumbar puncture/spinal catheterization.
14. Clinically significant abnormalities in coagulation parameters.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Part A and Part B cohorts B1-3 and B5-7: Healthy young male subjects, aged 18-50 years
  Part B cohort B4: Healthy male subjects and female subjects with non-childbearing potential aged 65 to 85 years
Enrollment: 32 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-09-09 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | Up to 12 days post initial dosing (Part A); Up to 19 days post initial dosing (Part B)
  Safety and tolerability of single or multiple ascending doses of ATH-1020 as measured by vital signs and clinical laboratory measurements.

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Cmax will be determined from all collected plasma samples from baseline through up to 48 hours post-dose.
  Cmax will be determined from all collected plasma samples from baseline through up to 48 hours post-dose.
Time to maximum observed plasma concentration (Tmax) | Samples collected pre-dose and at predetermined timepoints within 48 hours post-dose.
  Tmax will be determined from all collected plasma samples from baseline through up to 48 hours post-dose.
Plasma concentration at the end of the dosing interval (Ctrough) | Samples collected pre-dose and at predetermined timepoints within 24 hours post-dose.
  Ctrough will be determined from the last plasma sample prior to the following dose (cohort B only).
Area under the plasma concentration time curve (AUC) | Samples collected pre-dose and at predetermined timepoints within 48 hours post-dose.
  AUC will be determined from all collected plasma samples from baseline through up to 48 hours post-dose.
Half-life (t1/2) | Samples collected pre-dose and at predetermined timepoints within 48 hours post-dose.
  t1/2 will be determined from all collected plasma samples from baseline through up to 48 hours post-dose.
Amount of IMP excreted unchanged in the urine (Ae) | Samples collected pre-dose on Day 1 and predetermined timepoints on Day 1, 9, and 10, within 24 hours post-dose.
  Ae will be determined from all collected urine samples from baseline through up to 24 hours post-dose (cohort B1-4 only).

CONTACTS AND LOCATIONS:
Locations (1):
- Biotrial, Inc., Newark, New Jersey, United States